CLINICAL TRIAL: NCT04476472
Title: Evaluating the Safety and Effectiveness of the Omnipod Horizon™ Automated Glucose Control System in Children With Type 1 Diabetes Aged 2.0-5.9 Years: Preschool Cohort
Brief Title: Omnipod Horizon™ Automated Glucose Control System Preschool Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Horizon™ Preschool Cohort
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D; Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: single-arm, multi-center, prospective clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): All subjects wearing the Omnipod Horizon™ Automated Glucose Control System using the closed-loop algorithm.
  Interventions: Device: Omnipod Horizon™ Automated Glucose Control System

INTERVENTIONS:
Device: Omnipod Horizon™ Automated Glucose Control System — The Omnipod Horizon™ Automated Glucose Control System will provide automated insulin delivery.

SUMMARY:
Subjects will undergo a 14-day outpatient, standard therapy phase during which sensor and insulin data will be collected. This will be followed by a 94-day (13-week) hybrid closed-loop phase conducted in an outpatient setting, and an optional 12-month extension phase.

DETAILED DESCRIPTION:
The study schedule will consist of a standard therapy data collection phase followed by a hybrid closed-loop phase.

Subjects will undergo a 14-day outpatient, standard therapy phase during which sensor and insulin data will be collected. Subjects, or their caregivers, will manage their diabetes at home per their usual routine using the study continuous glucose monitoring system (CGM) and remain on current multiple daily injections (MDI) or pump therapy. This will be followed by a 94-day (13-week) hybrid closed-loop phase, conducted in an outpatient setting where subjects, or their caregivers, will manage their diabetes at home using the Omnipod Horizon™ Automated Glucose Control System. After completing the 94-day hybrid closed-loop phase, subjects will have the option to continue using the system for an additional 12 months.

During the hybrid closed-loop phase, a subset of subjects will participate in 2-days of supervised meal and exercise challenges.

The hybrid closed-loop phase will begin on Study Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 2.0-5.9 years
2. Living with parent/legal guardian
3. Diagnosed with type 1 diabetes. Diagnosis is based on investigator's clinical judgment
4. Deemed appropriate for pump therapy per investigator's assessment taking into account previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
5. Investigator has confidence that the subject and/or parent/guardian/caregiver can successfully operate all study devices and is capable of adhering to the protocol
6. Willing to use only the following types of insulin during the study: Humalog, Novolog, Admelog or Apidra during the study
7. Willing to wear the system continuously throughout the study
8. Willing to participate in challenges for 2 consecutive days, consisting of a minimum of 3 hours of activity per day and dietary challenge by reducing the number of carbohydrates entered for a given meal by 50%
9. A1C <10% at screening visit
10. Subject and/or parent/guardian must be willing to use the Dexcom App on the Omnipod Horizon™ PDM as the sole source of Dexcom data (with the exception of the Dexcom Follow App) during the hybrid closed-loop phase
11. Subject and/or parent/guardian is able to read and speak English fluently
12. Has a parent/legal guardian willing and able to sign the ICF.

Exclusion Criteria:

1. A medical condition, which in the opinion of the investigator, would put the subject at an unacceptable safety risk
2. History of severe hypoglycemia in the past 6 months
3. History of DKA in the past 6 months, unrelated to an intercurrent illness, infusion set failure or initial diagnosis
4. Diagnosed with sickle cell disease
5. Diagnosed with hemophilia or any other bleeding disorders
6. Plans to receive blood transfusion over the course of the study
7. Clinical evidence of acute or chronic kidney disease (e.g. estimated GFR < 45) or currently on hemodialysis
8. History of adrenal insufficiency
9. Has taken oral or injectable steroids within the past 8-weeks or plans to take oral or injectable steroids during the course of the study
10. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
11. Plans to use insulin other than U-100 insulin intended for use in the study device during the course of the study
12. Use of non-insulin anti-diabetic medication other than metformin (e.g. GLP1 agonist, SGLT2 inhibitor, DPP-4 inhibitor, pramlintide)
13. Thyroid Stimulating Hormone (TSH) is outside of normal range with clinical signs of hypothyroidism or hyperthyroidism
14. Currently participating or plans to participate in another clinical study using an investigational drug or device other than the Omnipod Horizon™ Automated Glucose Control System during this study period
15. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Study Chair — Stanford School of Medicine; Sue Brown, MD, Study Chair — University of Virginia
Locations (10):
- United States (10):
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Atlanta Diabetes, Atlanta, Georgia
  - Joslin Diabetes Center, Boston, Massachusetts
  - International Diabetes Center, Saint Louis Park, Minnesota
  - SUNY Syracuse, Syracuse, New York
  - University Hospitals Cleveland, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeSalvo DJ, Bode BW, Forlenza GP, Laffel LM, Buckingham BA, Criego AB, Schoelwer M, MacLeish SA, Sherr JL, Hansen DW, Ly TT. Glycemic Outcomes Persist for up to 2 Years in Very Young Children with the Omnipod(R) 5 Automated Insulin Delivery System. Diabetes Technol Ther. 2024 Jun;26(6):383-393. doi: 10.1089/dia.2023.0506. Epub 2024 Feb 21. PMID 38277156
- [Derived] Sherr JL, Bode BW, Forlenza GP, Laffel LM, Schoelwer MJ, Buckingham BA, Criego AB, DeSalvo DJ, MacLeish SA, Hansen DW, Ly TT; Omnipod 5 in Preschoolers Study Group:; Sherr JL, Weyman K, Tichy E, VanName M, Brei M, Zgorski M, Steffen A, Carria L, Bode BW, Busby A, Forlenza GP, Wadwa RP, Slover R, Cobry E, Messer L, Laffel LM, Isganaitis E, Ambler-Osborn L, Freiner E, Turcotte C, Volkening L, Schoelwer M, Brown SA, Krauthause K, Emory E, Oliveri M, Buckingham BA, Ekhlaspour L, Kingman R, Criego AB, Schwartz BL, Gandrud LM, Grieme A, Hyatt J, DeSalvo DJ, McKay S, DeLaO K, Villegas C, MacLeish SA, Wood JR, Kaminski BA, Casey T, Campbell W, Behm K, Adams R, Hansen DW, Stone SL, Bzdick S, Bulger J, Agostini L, Doolittle S, Kivilaid K, Kleve K, Ly TT, Dumais B, Vienneau T, Huyett LM, Lee JB, O'Connor J, Benjamin E. Safety and Glycemic Outcomes With a Tubeless Automated Insulin Delivery System in Very Young Children With Type 1 Diabetes: A Single-Arm Multicenter Clinical Trial. Diabetes Care. 2022 Aug 1;45(8):1907-1910. doi: 10.2337/dc21-2359. PMID 35678724

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Measure Description: Several participants identified as more than one race. Therefore, the sum of participants in this Baseline Measure will not be equal to the overall number of baseline participants.
  Participants
    American Indian or Alaska Native | 0
    Asian | 5
    Black or African American | 7
    Native Hawaiian or Other Pacific Islander | 0
    White | 72
    Other | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 16.7 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Severe Hypoglycemia (Events Per Person Months)
Description: Number of severe hypoglycemia events reported in "events per person months" units.
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (450 days)
Measure: Number; unit: events per person months
Arm/Group | Treatment
Number analyzed (Participants) | 80
events per person months
  Phase 2 | 0
  Phase 3 | 0.0007

2. Primary Outcome: Incidence Rate of Diabetic Ketoacidosis (DKA) (Events Per Person Months)
Description: Number of DKA events reported in "events per person months" units.
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (450 days)
Measure: Number; unit: events per person months
Arm/Group | Treatment
Number analyzed (Participants) | 80
events per person months
  Phase 2 | 0
  Phase 3 | 0.0007

3. Primary Outcome: Glycated Hemoglobin (A1C)
Description: Measures device effectiveness
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (180 days, 270 days, 360 days, and 450 days) compared to baseline
Measure: Mean (Standard Deviation); unit: percent A1C
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent A1C
  Baseline | 7.4 (1.0)
  V13 | 6.9 (0.7)
  V16 | 7.0 (0.7)
  V19 | 7.1 (0.7)
  V21 | 6.9 (0.7)
  V23 | 7.0 (0.7)

4. Primary Outcome: Time in Range 70-180 mg/dL
Description: Measures device effectiveness
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (450 days) compared to Phase 1 standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: percent time in range
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent time in range
  Day Time ST | 56.9 (15.2)
  Day Time Phase 2 | 63.7 (9.7)
  Day Time Phase 3 | 63.5 (9.8)
  Night Time ST | 58.2 (18.7)
  Night Time Phase 2 | 81.0 (10.0)
  Night Time Phase 3 | 78.2 (10.4)
  Overall ST | 57.2 (15.3)
  Overall Phase 2 | 68.1 (9.0)
  Overall Phase 3 | 67.2 (9.3)

5. Secondary Outcome: Glycated Hemoglobin (A1C)
Description: Measures device effectiveness
Time Frame: Hybrid closed-loop (94 days, 180 days, 270 days, and 450 days) compared to baseline
Measure: Mean (Standard Deviation); unit: percent A1C
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent A1C
  Baseline | 7.4 (1.0)
  V13 | 6.9 (0.7)
  V16 | 7.0 (0.7)
  V19 | 7.1 (0.7)
  V21 | 6.9 (0.7)
  V23 | 7.0 (0.7)

6. Secondary Outcome: Percent of Time in Range 70-140 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (450 days) compared to Phase 1 standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: percent time in range
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent time in range
  Day Time ST | 36.2 (13.2)
  Day Time Phase 2 | 41.3 (9.4)
  Day Time Phase 3 | 41.2 (9.8)
  Night Time ST | 36.7 (16.9)
  Night Time Phase 2 | 57.7 (13.7)
  Night Time Phase 3 | 53.9 (13.1)
  Overall ST | 36.3 (13.4)
  Overall Phase 2 | 45.4 (9.7)
  Overall Phase 3 | 44.4 (10.0)

7. Secondary Outcome: Percent of Time > 180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of time
  Day Time ST | 39.7 (16.6)
  Day Time Phase 2 | 33.7 (10.7)
  Day Time Phase 3 | 33.7 (10.8)
  Night Time ST | 38.4 (20.1)
  Night Time Phase 2 | 16.9 (10.3)
  Night Time Phase 3 | 19.7 (10.6)
  Overall ST | 39.4 (16.7)
  Overall Phase 2 | 29.5 (9.8)
  Overall Phase 3 | 30.2 (10.1)

8. Secondary Outcome: Percent of Time ≥ 250 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of time
  Day Time ST | 15.4 (12.7)
  Day Time Phase 2 | 11.0 (6.6)
  Day Time Phase 3 | 11.5 (6.9)
  Night Time ST | 13.0 (13.2)
  Night Time Phase 2 | 3.9 (3.9)
  Night Time Phase 3 | 5.1 (4.6)
  Overall ST | 14.8 (12.1)
  Overall Phase 2 | 9.2 (5.6)
  Overall Phase 3 | 9.9 (6.0)

9. Secondary Outcome: Percent of Time ≥ 300 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of time
  Day Time ST | 6.5 (8.0)
  Day Time Phase 2 | 3.9 (3.4)
  Day Time Phase 3 | 4.4 (3.8)
  Night Time ST | 4.3 (6.7)
  Night Time Phase 2 | 1.2 (1.6)
  Night Time Phase 3 | 1.8 (2.1)
  Overall ST | 6.0 (7.3)
  Overall Phase 2 | 3.2 (2.8)
  Overall Phase 3 | 3.7 (3.2)

10. Secondary Outcome: Percent of Time < 70 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of time
  Day Time ST | 3.44 (3.85)
  Day Time Phase 2 | 2.57 (1.99)
  Day Time Phase 3 | 2.79 (1.98)
  Night Time ST | 3.41 (4.79)
  Night Time Phase 2 | 2.13 (1.94)
  Night Time Phase 3 | 2.06 (1.70)
  Overall ST | 3.43 (3.87)
  Overall Phase 2 | 2.46 (1.83)
  Overall Phase 3 | 2.61 (1.82)

11. Secondary Outcome: Percent of Time < 54 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of time
  Day Time ST | 0.80 (1.67)
  Day Time Phase 2 | 0.50 (0.61)
  Day Time Phase 3 | 0.59 (0.63)
  Night Time ST | 0.85 (1.94)
  Night Time Phase 2 | 0.39 (0.53)
  Night Time Phase 3 | 0.49 (0.63)
  Overall ST | 0.81 (1.68)
  Overall Phase 2 | 0.47 (0.54)
  Overall Phase 3 | 0.57 (0.60)

12. Secondary Outcome: Mean Glucose
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 80
mg/dL
  Day Time ST | 172.2 (31.3)
  Day Time Phase 2 | 163.0 (18.3)
  Day Time Phase 3 | 163.6 (19.3)
  Night Time ST | 168.1 (33.3)
  Night Time Phase 2 | 140.7 (16.4)
  Night Time Phase 3 | 145.7 (16.9)
  Overall ST | 171.1 (30.5)
  Overall Phase 2 | 157.4 (16.8)
  Overall Phase 3 | 159.1 (17.9)

13. Secondary Outcome: Standard Deviation
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the standard deviation (SD)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 80
mg/dL
  Day Time ST | 66.1 (13.7)
  Day Time Phase 2 | 62.2 (10.5)
  Day Time Phase 3 | 63.4 (11.3)
  Night Time ST | 58.0 (14.0)
  Night Time Phase 2 | 45.5 (10.8)
  Night Time Phase 3 | 48.8 (11.7)
  Overall ST | 64.9 (13.4)
  Overall Phase 2 | 59.6 (10.3)
  Overall Phase 3 | 60.9 (11.1)

14. Secondary Outcome: Coefficient of Variation
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent coefficient of variation
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent coefficient of variation
  Day Time ST | 38.6 (5.7)
  Day Time Phase 2 | 38.0 (3.8)
  Day Time Phase 3 | 38.6 (3.7)
  Night Time ST | 34.7 (6.6)
  Night Time Phase 2 | 32.1 (5.2)
  Night Time Phase 3 | 33.2 (5.1)
  Overall ST | 38.1 (5.5)
  Overall Phase 2 | 37.7 (4.0)
  Overall Phase 3 | 38.1 (3.9)

15. Secondary Outcome: Percentage of Time in Hybrid Closed-loop as Proportion of Overall Device Usage Time
Description: Measure of system usage in Automated and Manual modes. Percentage of time in Automated and Manual mode do not add up to 100% due to missing data from participants not using the Omnipod 5 system (e.g., not wearing a Pod).
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 (450 days)
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of time
  Phase 2 Automated Mode | 96.8 (2.6)
  Phase 2 Manual Mode | 2.8 (2.5)
  Phase 3 Automated Mode | 95.5 (3.8)
  Phase 3 Manual Mode | 3.2 (3.2)

16. Secondary Outcome: Glucose Management Indicator (GMI)
Description: Glucose Management Indicator (%) approximates the laboratory hemoglobin A1c (%) expected based on average glucose readings from continuous glucose monitors from the last 14 days or more.
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (450 days) compared to the Phase 1 standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: percent of gmi
Arm/Group | Treatment
Number analyzed (Participants) | 80
percent of gmi
  Day Time ST | 7.43 (0.75)
  Day Time Phase 2 | 7.21 (0.44)
  Day Time Phase 3 | 7.22 (0.46)
  Night Time ST | 7.33 (0.80)
  Night Time Phase 2 | 6.68 (0.39)
  Night Time Phase 3 | 6.79 (0.40)
  Overall ST | 7.40 (0.73)
  Overall Phase 2 | 7.08 (0.40)
  Overall Phase 3 | 7.12 (0.43)

17. Secondary Outcome: Total Daily Insulin (TDI) (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Treatment
Number analyzed (Participants) | 80
units
  ST | 13.7 (4.4)
  Phase 2 | 14.1 (4.0)
  Phase 3 | 16.4 (4.5)

18. Secondary Outcome: Total Daily Insulin (TDI) (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Treatment
Number analyzed (Participants) | 80
units/kg
  ST | 0.69 (0.18)
  Phase 2 | 0.71 (0.15)
  Phase 3 | 0.80 (0.17)

19. Secondary Outcome: Total Daily Basal Insulin (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Treatment
Number analyzed (Participants) | 80
units
  ST | 5.6 (2.5)
  Phase 2 | 6.4 (2.4)
  Phase 3 | 7.7 (2.8)

20. Secondary Outcome: Total Daily Basal Insulin (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Treatment
Number analyzed (Participants) | 80
units/kg
  ST | 0.28 (0.12)
  Phase 2 | 0.32 (0.10)
  Phase 3 | 0.38 (0.11)

21. Secondary Outcome: Total Daily Bolus Insulin (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Treatment
Number analyzed (Participants) | 80
units
  ST | 8.1 (3.3)
  Phase 2 | 7.7 (2.3)
  Phase 3 | 8.7 (2.5)

22. Secondary Outcome: Total Daily Bolus Insulin (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 16
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Treatment
Number analyzed (Participants) | 80
units/kg
  ST | 0.41 (0.15)
  Phase 2 | 0.39 (0.10)
  Phase 3 | 0.42 (0.11)

23. Secondary Outcome: Body Mass Index (BMI) (kg/m^2)
Description: Measure of change in weight
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (450 days) compared to baseline
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment
Number analyzed (Participants) | 80
kg/m^2
  Baseline | 16.7 (1.5)
  V13 | 16.7 (1.4)
  V23 | 16.9 (2.3)

ADVERSE EVENTS:
Time Frame: First day of standard therapy phase until participant's participation in study ended, an average of 15 weeks.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 4/80
Other Adverse Events (participants affected / at risk) | 51/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=80)
Severe hypoglycemia (Endocrine disorders) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1)
Prolonged Hyperglycemia (Endocrine disorders) | 1 (1)
Other (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=80)
Hypoglycemia (Endocrine disorders) | 2 (2)
Prolonged Hyperglycemia (Endocrine disorders) | 26 (51)
Hyperglycemia (Endocrine disorders) | 3 (3)
Other (Endocrine disorders) | 36 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT04476472/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT04476472/SAP_001.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT04476472/ICF_002.pdf